CLINICAL TRIAL: NCT06756802
Title: Reproductive Health in Breast Cancer Survivor
Acronym: ISIS
Status: Active, not recruiting | Type: Observational
Sponsor: Institut Cancerologie de l'Ouest (Other)
Collaborators: UNICANCER (Other)
Responsible Party: Sponsor
Other Study IDs: ICO-2021-41
Record Dates: First submitted 2024-12-04; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer
Keywords: breast cancer; health reproductive; fertility
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Exposed cohort: Patients in ConSoRe data with a diagnosis of stage 1 to 3 breast cancer between 01/01/2010 and 31/12/2018.
- Non-exposed cohort: Women present in the SNDS data, without a diagnosis of breast cancer, born between 01/01/1970 and 31/12/2000.
- Cohort associated with the exposed cohort: Children of included patients born after diagnosis of breast cancer.

SUMMARY:
With the age of first pregnancy increasing (average age of mother at childbirth: 31.0 in 2022), and the incidence of breast cancer increasing in young women (+2.1% per year according to some registries, more and more women will develop breast cancer before they have a child. FP must be offered to all women under 40 who are going to receive potentially gonadotoxic treatment (French bioethics law of 06/08/04, revised on 07/07/2011). It therefore seems appropriate to collect data from patients aged between 18 and 40 at diagnosis (previous fertility, fertility preservation before chemotherapy). Furthermore, the theoretical risk of pregnancy persists until the menopause. For the study of contraception, patients aged up to 50 at diagnosis will therefore be included. In view of the EMA's recent warning on the genotoxic risk of tamoxifen, the investigator feel that it would be relevant to collect data on the health status of newborns born after breast cancer (three compulsory medical examinations in the first month of life to detect any malformative pathologies).

A better understanding of these issues would enable national and even international recommendations to be updated, patients to be better informed and the long-term consequences on fertility to be better managed.

DETAILED DESCRIPTION:
The impact of cancer treatments on reproductive life and the health of unborn children is a major concern for young patients diagnosed and treated for cancer.

The information gathered by this project will make it possible to provide clearer and more accurate information to patients about the consequences of cancer therapies on their reproductive lives. In addition, the investigator hope to be able to reassure doctors about the use of fertility preservation before breast cancer and MPA after breast cancer, and to have arguments for fertility preservation and MPA to be offered more systematically to patients.

Answering such questions in prospective trials would require a long follow-up period and the inclusion of a very large number of patients. The creation of a multicentre retrospective database could provide answers to a large number of questions about the impact of anti-cancer therapies on reproductive life in the management of female breast cancer. In addition, to limit the risk of bias, these data will be compared with those of a population of women of the same age without breast cancer.

ELIGIBILITY:
Exposed cohort (Breast cancer patient)

Inclusion Criteria:

* Patients aged between 18 and 50 at the time of diagnosis of breast cancer
* Diagnosed with stage 1 to 3 breast cancer between 01/01/2010 and 31/12/2018
* Patients treated in one of the identified ConSoRe partner centres (CLB, ICO, COL, IC)

Exclusion Criteria:

* Diagnosis of metastatic breast cancer (stage 4)
* Patients opposed to the use of their data for research purposes

Unexposed cohort (data from the SNDS) :

Population derived from the SNDS, among women not diagnosed with breast cancer, of the same ages (same year of birth) and the same geographical area (same département of residence) as the exposed population.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women with Breast cancer / Women not diagnosed with breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 22000 (Estimated)
Dates: Start 2024-07-11 (Actual); Primary Completion 2029-07-11 (Estimated); Study Completion 2029-07-11 (Estimated)

PRIMARY OUTCOMES:
to describe pregnancies (number, origin and outcome) after stage 1 to 3 breast cancer in women aged 18 to 40 at diagnosis, according to age at diagnosis and treatment received. | 4 years
  Number of spontaneous and MPA pregnancies, with viable child or not, after stage 1 to 3 breast cancer in women aged 18 to 40 at diagnosis, according to age at diagnosis and treatments received.

SECONDARY OUTCOMES:
a) Compare the pregnancy rate after breast cancer, for patients aged 18 to 40 at the time of diagnosis of breast cancer, with the pregnancy rate in a sample of women without breast cancer from the general population, overall and, for patients, by sub-gro | 4 years
  Pregnancy rates, as well as all the criteria mentioned in the primary endpoint, will be compared between patients with stage 1 to 3 breast cancer aged 18 to 40 at the time of diagnosis and women without breast cancer from the SNDS. Subpopulations according to treatment will concern only the exposed population.
b) To describe the use of fertility preservation before chemotherapy: oncofertility consultation, preservation techniques for patients aged between 18 and 40 at the time of diagnosis of breast cancer. | 4 years
  Number of oncofertility consultations and number of fertility preservation acts for each preservation technique, for women with stage 1 to 3 breast cancer, aged 18 to 40 at diagnosis.
c) Describe the link between recourse to MAP after cancer and the risk of recurrence, for patients aged between 18 and 40 at the time of diagnosis of breast cancer. | 4 years
  Relapse-free survival for women with stage 1 to 3 breast cancer, aged 18 to 40 at diagnosis according to the use of MAP method.
d) To describe the risk of breast cancer recurrence according to the time between stopping and restarting tamoxifen, for patients aged 18 to 40 at the time of diagnosis of breast cancer. | 4 years
  The risk of breast cancer recurrence will be assessed by recurrence-free survival according to the duration between stopping and restarting tamoxifen, for patients aged 18 to 40 at the time of breast cancer diagnosis.
e) To describe fetal malformations and perinatal pathologies in children born according to the duration of tamoxifen discontinuation (3 to 9 months vs. > 9 months), for patients aged 18 to 40 years at the time of breast cancer diagnosis. | 4 years
  Fetal malformations and perinatal pathologies of the children born will be evaluated by the rates of FCS, fetal malformations, IMG, fetal deaths in utero, neonatal deaths according to the duration of tamoxifen discontinuation (between 3 and 9 months vs. > 9 months), for patients aged 18 to 40 years at the time of breast cancer diagnosis.
f) To describe fetal malformations and perinatal pathologies in children born after tamoxifen was stopped 3 to 9 months before the start of pregnancy and after no tamoxifen was taken, in patients aged 18 to 40 at the time of diagnosis of breast cancer. | 4 years
  Fetal malformations and perinatal pathologies of the children born will be evaluated by the rates of FCS, fetal malformations, IMG, fetal deaths in utero, neonatal deaths, for patients who received tamoxifen and stopped between 3 and 9 months before pregnancy, and for patients who did not receive tamoxifen, among patients aged 18 to 40 years at the time of breast cancer diagnosis.
g) To describe the care pathway for patients aged between 18 and 50 at the time of diagnosis of breast cancer | 4 years
  Time between the diagnostic and, on one hand, first medical gesture, and the other hand, oncogenetic consultation, for women with stage 1 to 3 breast cancer, aged 18 to 50 at diagnosis
h) To describe contraception and the rate of abortion during and after treatment for breast cancer in patients aged between 18 and 50 at the time of their diagnosis. | 4 years
  Number of women using a contraceptive method and number of unwanted prenancies, for women with stage 1 to 3 breast cancer, aged 18 to 40 at diagnosis, during and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Aliette DEZELLUS, MD, Principal Investigator — INSTITUT DE CANCEROLOGIE DE L'OUEST; Marie ROBERT, MD, Principal Investigator — INSTITUT DE CANCERORLOGIE DE L'OUEST
Locations (4):
- France (4):
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Institut Curie, Paris
  - Institut de Cancerologie de L'Ouest, Saint-Herblain

IPD SHARING:
Plan to Share IPD: Yes
The base will be added to the HDH catalogue
Supporting Information: CSR
Time Frame: Unknowed